CLINICAL TRIAL: NCT04397458
Title: Rescue Quadratus Lumborum Blocks for Post-cesarean Pain
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: COVID-19 pandemic and competing study that took precedence
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Maya Suresh, Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC-MS-20-0124
Record Dates: First submitted 2020-05-04; First posted 2020-05-21 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: Morphine; Analgesics; Analgesics, Opioid; Peripheral Nervous System Agents
Keywords: quadratus lumborum block; bupivacaine; cesarean delivery; c-section; intrathecal morphine; post-operative pain; post-cesarean analgesia
MeSH Terms: conditions — Pain, Postoperative | interventions — Sodium Chloride; Bupivacaine; Dexamethasone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sham Control (Sham Comparator): 20 milliliters (mL) 0.9% saline on each side
  Interventions: Drug: Saline
- Quadratus Lumborum Block (Experimental): 20 mL solution with 0.25% bupivacaine (50 milligrams (mg)) and 3mg preservative-free dexamethasone on each side
  Interventions: Drug: Bupivacaine; Drug: Dexamethasone

INTERVENTIONS:
Drug: Saline — 0.9% saline on each side
  Arms: Sham Control
Drug: Bupivacaine — 0.25% bupivacaine (50mg) on each side
  Arms: Quadratus Lumborum Block
Drug: Dexamethasone — 3mg preservative-free dexamethasone on each side
  Arms: Quadratus Lumborum Block

SUMMARY:
The purpose of this study is to assess whether quadratus lumborum (QL) block performed 1 day after cesarean delivery will provide supplemental post-cesarean analgesia and reduce opioid requirements.

ELIGIBILITY:
Inclusion Criteria:

* elective or non-elective cesarean delivery on prior day
* pain scores >5/10

Exclusion Criteria:

* BMI >40
* obstructive sleep apnea
* drug abuse
* chronic pain
* chronic opioid use
* abdominal surgeries other than cesarean delivery
* contraindications to neuraxial or regional anesthesia
* received general anesthesia or did not receive neuraxial morphine for cesarean delivery

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Total opioid consumption | 48 hours after intervention

SECONDARY OUTCOMES:
Amount of opioids used | at the time of intervention (one day following cesarean delivery)
Amount of opioids used | 6 hours after intervention
Amount of opioids used | 12 hours after intervention
Amount of opioids used | 24 hours after intervention
Amount of opioids used | 48 hours after intervention
Time from quadratus lumborum block until first opioid request | from time of intervention until time of first opioid request (up to 48 hours)
Pain as measured by an 11-point verbal pain score (at rest) | at the time of intervention (one day following cesarean delivery)
  The 11-point verbal pain score ranges from 0-10, with a higher number indicating worse pain.
Pain as measured by an 11-point verbal pain score (with movement) | at the time of intervention (one day following cesarean delivery)
  The 11-point verbal pain score ranges from 0-10, with a higher number indicating worse pain.
Pain as measured by an 11-point verbal pain score (at rest) | 6 hours after intervention
  The 11-point verbal pain score ranges from 0-10, with a higher number indicating worse pain.
Pain as measured by an 11-point verbal pain score (with movement) | 6 hours after intervention
  The 11-point verbal pain score ranges from 0-10, with a higher number indicating worse pain.
Pain as measured by an 11-point verbal pain score (at rest) | 12 hours after intervention
  The 11-point verbal pain score ranges from 0-10, with a higher number indicating worse pain.
Pain as measured by an 11-point verbal pain score (with movement) | 12 hours after intervention
  The 11-point verbal pain score ranges from 0-10, with a higher number indicating worse pain.
Pain as measured by an 11-point verbal pain score (at rest) | 24 hours after intervention
  The 11-point verbal pain score ranges from 0-10, with a higher number indicating worse pain.
Pain as measured by an 11-point verbal pain score (with movement) | 24 hours after intervention
  The 11-point verbal pain score ranges from 0-10, with a higher number indicating worse pain.
Pain as measured by an 11-point verbal pain score (at rest) | 48 hours after intervention
  The 11-point verbal pain score ranges from 0-10, with a higher number indicating worse pain.
Pain as measured by an 11-point verbal pain score (with movement) | 48 hours after intervention
  The 11-point verbal pain score ranges from 0-10, with a higher number indicating worse pain.
Nausea as measured by a 3-point scale | at the time of intervention (one day following cesarean delivery)
  This is measured categorically as none, mild, or moderate-severe.
Nausea as measured by a 3-point scale | 6 hours after intervention
  This is measured categorically as none, mild, or moderate-severe.
Nausea as measured by a 3-point scale | 12 hours after intervention
  This is measured categorically as none, mild, or moderate-severe.
Nausea, pruritus and sedation as measured by a 3-point scale | 24 hours after intervention
  This is measured categorically as none, mild, or moderate-severe.
Nausea as measured by a 3-point scale | 48 hours after intervention
  This is measured categorically as none, mild, or moderate-severe.
Pruritus as measured by a 3-point scale | at the time of intervention (one day following cesarean delivery)
  This is measured categorically as none, mild, or moderate-severe.
Pruritus as measured by a 3-point scale | 6 hours after intervention
  This is measured categorically as none, mild, or moderate-severe.
Pruritus as measured by a 3-point scale | 12 hours after intervention
  This is measured categorically as none, mild, or moderate-severe.
Pruritus as measured by a 3-point scale | 24 hours after intervention
  This is measured categorically as none, mild, or moderate-severe.
Pruritus as measured by a 3-point scale | 48 hours after intervention
  This is measured categorically as none, mild, or moderate-severe.
Sedation as measured by a 3-point scale | at the time of intervention (one day following cesarean delivery)
  This is measured categorically as none, mild, or moderate-severe.
Sedation as measured by a 3-point scale | 6 hours after intervention
  This is measured categorically as none, mild, or moderate-severe.
Sedation as measured by a 3-point scale | 12 hours after intervention
  This is measured categorically as none, mild, or moderate-severe.
Sedation as measured by a 3-point scale | 24 hours after intervention
  This is measured categorically as none, mild, or moderate-severe.
Sedation as measured by a 3-point scale | 48 hours after intervention
  This is measured categorically as none, mild, or moderate-severe.
Patient satisfaction as measured by the 5-point Likert scale | 48 hours after intervention
  The 5-point scale ranges from extremely satisfied to not satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Linden Lee, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No